CLINICAL TRIAL: NCT07173543
Title: Intermittent Hypoxia Training and Cerebrovascular Health in Older Adults With Type 2 Diabetes
Brief Title: IH, Brain Health, and T2D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Darren P Casey (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Sponsor-Investigator, Darren P Casey, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 202505661
Record Dates: First submitted 2025-09-02; First posted 2025-09-15 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes; Aging
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intermittent Hypoxia 1 (Experimental): Participants will receive intermittent hypoxia (5 cycles of normoxia/hypoxia over 50 minutes).
  Interventions: Other: Intermittent Hypoxia 1 (IH1)
- Normoxia (Sham Comparator): Participants will receive normoxia over 50 minutes.
  Interventions: Other: SHAM - normoxia
- Intermittent Hypoxia 2 (Experimental): Participants will receive intermittent hypoxia (5 cycles of normoxia/hypoxia over 50 minutes).
  Interventions: Other: Intermittent Hypoxia 2 (IH2)

INTERVENTIONS:
Other: Intermittent Hypoxia 1 (IH1) — Intermittent Hypoxia 1 (IH1): 5 cycles of normoxia (4 minutes)/hypoxia (6 minutes) per session. 3 sessions per week for 8 weeks
  Arms: Intermittent Hypoxia 1
Other: Intermittent Hypoxia 2 (IH2) — Intermittent Hypoxia 1 (IH2): 5 cycles of normoxia (4 minutes)/hypoxia (6 minutes) per session. 3 sessions per week for 4 weeks
  Arms: Intermittent Hypoxia 2
Other: SHAM - normoxia — Participants will receive normoxia (no hypoxia) over 50 minutes.
  Arms: Normoxia

SUMMARY:
The purpose of this study is to use a randomized, placebo-controlled study design to rigorously examine the therapeutic potential of intermittent hypoxia (IH) for improving cerebrovascular health in older adults with and without type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
Aging is considered a major risk factor for the development of various cardio- and cerebrovascular related diseases, with vascular endothelial dysfunction representing one of the earliest vascular complications. Age-related cerebrovascular endothelial dysfunction contributes to a progressive decrease in cerebral blood flow, which is associated with lower measures of cognitive function, including information-processing speed, executive function, and global cognition in older adults. Similar to aging, type 2 diabetes mellitus (T2DM) also negatively impacts vascular endothelial function. There is a large body of evidence that clearly demonstrates there is an interplay between aging and T2DM and that the presence of both risk factors together promotes greater endothelial dysfunction than that of either condition alone. In this context, certain measures of cerebral blood flow are reduced to a greater extent in older individuals with T2DM compared to those without. Moreover, the exaggerated cerebral perfusion deficits frequently observed among older adults with T2DM are linked to cognitive decrements. To this point, the rate of cognitive decline due to aging is increased 1.5 to 2.0-fold in individuals with T2DM. Taken together, older adults with T2DM are at greater risk for developing dementia and Alzheimer's disease when compared age-matched controls.

Exploration of non-pharmacological therapies for the improvement of cerebrovascular health and cognition have become more common over the past decade. Intermittent hypoxia (IH) is a therapeutic intervention that combines multiple, brief (~1-10 minutes) episodes of moderate hypoxia, interspersed with episodes of normoxia. In preclinical and human studies, repeated bouts of IH improve measures of respiratory, autonomic, cardio-, and cerebrovascular health. The investigators previously demonstrated that cerebral blood flow is increased with each episode of hypoxia and a single session of IH improves nitic oxide (NO) mediated endothelial function in the internal carotid artery (ICA; major supplier of overall brain blood flow) of young adults. While cerebral blood flow is also augmented during a single session of IH in older adults, the magnitude of change appears to be less, which might suggest older adults with and without T2DM may need repeated sessions of IH for improvements in cerebrovascular health to occur. The investigator's central hypothesis is that experimental use of IH will effectively and progressively improve cerebrovascular health and cognition in older adults with T2DM. Specifically, the investigators will evaluate the interplay between aging and T2DM and how it influences cerebral endothelial function as well as the cerebrovascular responses to IH (Aim 1) and test the effectiveness of IH training for the improvement of cerebrovascular health in older adults living with diabetes (Aim 2). Collectively, the proposed studies will provide 1) novel understanding of cerebrovascular function in older adults with and without T2DM, and 2) important insight into the therapeutic potential of IH for improving cerebrovascular health and cognition in older adults living with T2DM.

ELIGIBILITY:
For 30 patients with documented Type 2 diabetes

Inclusion Criteria:

* Willing and able to provide written, signed informed consent after the nature of the study has been explained, and prior to any research-related procedures.
* Age is > or = 60 and < or = 85 years of age
* Documented Type 2 diabetes
* Scoring 26 or higher on the MoCA test

Exclusion criteria:

* diagnosis of type 2 diabetes < 1 year prior to enrollment
* HbA1c <6.5% or >10.0%
* body mass index > 40 kg/m 2
* incident cardiovascular events in the last year (heart attack, stroke)
* symptomatic coronary artery disease and/or heart failure
* uncontrolled hypertension
* obstructive sleep apnea
* pulmonary disease
* dementia
* renal impairment with creatinine clearance (eGFR) of <60 ml/min
* smoking or history of smoking within past one year

  30 nondiabetic control subjects will also be studied.

Inclusion criteria:

* Willing and able to provide written, signed informed consent after the nature of the study has been explained, and prior to any research-related procedures.
* Age is > or = 60 and < or = 85 years of age
* Scoring 26 or higher on the MoCA test

Exclusion criteria:

* Diagnosis of diabetes (Type 1 or Type 2)
* body mass index > 40 kg/m2
* incident cardiovascular events in the last year (heart attack, stroke)
* symptomatic coronary artery disease and/or heart failure
* uncontrolled hypertension
* obstructive sleep apnea
* pulmonary disease
* dementia
* renal impairment with creatinine clearance (eGFR) of <60 ml/min
* smoking or history of smoking within past one year

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-22 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Internal Carotid Artery (ICA) shear-mediated dilation | Baseline and post 2-,4-,5-,6-, and 8-weeks
  ICA dilation (% change) will be determined using Doppler ultrasound in response to acute hypercapnia.
Cerebral blood flow responsiveness | Baseline and after 50 minutes of IH or SHAM
  Cerebral blood flow will be determined using Doppler ultrasound in response to acute hypoxia.
Cognitive function testing | Baseline and post 4- and 8-weeks
  Working memory will be assessed using a facial recognition n-back task test

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa, Iowa City, Iowa, United States